## CONSENT BY PATIENT FOR CLINICAL RESEARCH

Version No.: 1

| Version Date: 1st April 2020 |
|---|
| I, |
| of |
| <u>Title of Study:</u> The Feasibility and Impact of a Home-based NMES program on Post-stroke Lower Limb Spasticity. |
| the nature and purpose of which has been explained to me by Dr |
| (Name & Designation of Doctor) |
| and interpreted by(Name & Designation of Interpreter) |
| to the best of his/her ability inlanguage/dialect. |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per patient information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent of my own free will to participate in the clinical research specified above. |
| I understand that I can withdraw from this clinical research at any time without assigning any reason whatsoever and in such a situation shall not be denied the benefits of usual treatment by the attending doctors. |
| Date: |
| IN THE PRESENCE OF |
| Name) |
| Identity Card No |
| (Witness for Signature of Patient) Designation) |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research. |
| Date |
| CONSENT BY PATIENT R.N. |

Name

Sex Age Unit

FOR CLINICAL RESEARCH

BK-MIS-1117-E02